CLINICAL TRIAL: NCT02615847
Title: A Phase II, Open Label, Single Center Trial to Study the Safety and Tolerability of Memantin Mepha® as Supportive Long Term Treatment in Symptomatic Sickle Cell Disease
Brief Title: Clinical Trial to Study the Safety and Tolerability of Memantin Mepha® in Sickle Cell Disease Patients
Acronym: MemSID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HbSS-MemSID
Record Dates: First submitted 2015-09-07; First posted 2015-11-26 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantin arm (Experimental): Memantinhydrochlorid, administered once per day during 12 month. Dosage is from 0-20 mg.
  Interventions: Drug: Memantinhydrochlorid

INTERVENTIONS:
Drug: Memantinhydrochlorid — Memantin Mepha® Lactabs (memantinehydrochlorid) will be provided as 5 mg, 10 mg, 15 mg and 20 mg tablets, packed in blister.
  The study drug will be taken once a day per os, during 12 month.
  Other Names: Memantin Mepha

SUMMARY:
Symptomatic sickle cell disease is worldwide the most frequent cause for hereditary hemolytic anemia with recurrent pain crisis. Hemolysis, vaso- occlusive and pain crises are hallmarks of this disease and are causative for an important socio-economic burden worldwide, especially in Africa.

Aside from allogenic stem cell transplantation, which is rarely available and very expensive, at present there is no curative treatment for patients with sickle cell disease (SCD). The current standard of care includes treatment with hydroxycarbamide and symptomatic care such as transfusions, antibiotic/analgesic treatment.

This study has the aim to study the safety and tolerability of Memantin in patients with sickle cell disease.

DETAILED DESCRIPTION:
During the study participants will be asked if medical occurrences (AEs) happened and laboratory analysis (haematology, coagulation, chemistry) and urine samples will be taken. In addition at each visit a physical examination and measurement of vital signs will be performed.

In addition the number of hospital days and emergency consultations, the impact on working ability (the number of days with inability to work, changes in iv%), the amount and type of analgesic medication, the amount of RBC transfusions, the number of days that antibiotics prescribed and haematology (at local and external laboratory) and chemistry laboratory parameters will be assessed. For the impact on work and social life a questionnaire of quality of life will be filled out monthly by the patient.

At screening and at the end of the study SCD specific assessments will be performed, which include cardiologic examination (ECG, ECHO), abdominal sonography, ophthalmological examination, lung function testing and neuroangiologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic sickle cell disease (HbSS or HbS/beta thalassemia)

  * Age 18 years or older
  * Able and willing to provide written informed consent and to comply with the study protocol procedures
  * Willing to use two effective methods of contraception during study treatment until 6 months after stop of study treatment. Effective contraception methods are considered oral, injectable, implantative contraceptives or intrauterine contraceptive devices combined with the use of condom.

Exclusion Criteria:

* History of transfusion during last three months before Screening

  * Patients with active bacterial, viral or fungal infection requiring systemic treatment
  * Patients with known infection with human immunodeficiency virus (HIV) of human T cell leukaemia virus 1 (HTLV-1)
  * Inadequate renal function: creatinine clearance < 30ml/min
  * Inadequate liver function: NCICTC Grade 3 liver function tests (AST, ALT > 5x upper limit of normal (ULN))
  * History of malignancy
  * Women who are pregnant or breast feeding
  * Previous known mental disorder or known family history of psychiatric diseases
  * Known epileptic disease
  * The receipt of any investigational product within 30 days prior to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03-31 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE version 4.0 | 14 month

SECONDARY OUTCOMES:
Haemoglobin in g/l | 38 month
  2 years before screening until end of study.
Erythrocytes in T/l | 38 month
  2 years before screening until end of study.
Reticulocytes in G/l | 38 month
  2 years before screening until end of study.
Haptoglobin in g/l | 38 month
  2 years before screening until end of study.
Billirubin in micmol/l | 38 month
  2 years before screening until end of study.
LDH (Lactat dehydrogenase) in U/l | 38 month
  2 years before screening until end of study.
Ferritin in micg/l | 38 month
  2 years before screening until end of study.
Transferrin saturation in % | 38 month
  2 years before screening until end of study.
Number of days in hospital | 38 month
  2 years before screening until end of study.
Number of days with inability to work | 38 month
  2 years before screening until end of study.
Number of transfusions | 38 month
  2 years before screening until end of study.
Number of days taken antibiotics | 38 month
  2 years before screening until end of study.
Amount of pain medication in mg or ml | 38 month
  2 years before screening until end of study.
Pain scale | 38 month
  Scores range from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Goede, MD, Study Chair — Universitätsspital Zürich
Locations (1):
- University Hospital Zürich, Zurich, Switzerland